CLINICAL TRIAL: NCT00964054
Title: Adapting Exercise Treatment for Depression to Adolescents: A Pilot Study
Brief Title: Depression Outcomes Study of Exercise
Acronym: DOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH082153 (NIH); MH082153; DSIR 84-CTS
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2012-04

CONDITIONS: Unipolar Depression
Keywords: adolescents; exercise; depression; dose response; pilot study
MeSH Terms: conditions — Depressive Disorder; Motor Activity; Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Public Health Dose of Exercise (PHD) (Experimental): 17.5 kcal per kilogram per week
  Interventions: Other: Public Health Dose of Exercise (PHD)
- Low Dose Exercise (LD) (Active Comparator): 7.0 kcal per kilogram per week
  Interventions: Other: Low Dose Exercise (LD)

INTERVENTIONS:
Other: Public Health Dose of Exercise (PHD) — 17.5 kcal per kilogram per week
  Other Names: Exercise; Physical Activity
  Arms: Public Health Dose of Exercise (PHD)
Other: Low Dose Exercise (LD) — 7.0 kcal per kilogram per week
  Other Names: Exercise; Physical Activity
  Arms: Low Dose Exercise (LD)

SUMMARY:
This pilot study may yield important research findings on how to adapt exercise treatment for depression among adolescents. Potential public health benefits from this study include a reduction of adolescent depression and problems associated with untreated depression in young adults including suicide, substance abuse, cigarette smoking, teen pregnancy, impaired psychosocial functioning and school failure. In addition, because this study prescribes physical activity as a treatment for depression, additional public health benefits may include a reduction in chronic diseases such as obesity, diabetes and heart disease, all of which are associated with sedentary behavior.

DETAILED DESCRIPTION:
Adolescent depression is a major public health problem in the United States and throughout the world. Major depressive disorder (MDD) in adolescence is common with point prevalence rates of 3% to 9%. In the U.S., it is estimated that by the time adolescents reach the age of 17, 14% will have experienced at least one episode of major depressive disorder. Effective treatments of adolescent depression are clearly needed despite the fact that in the past 10-15 years, there has been a dramatic increase in studies of the efficacy of medications, primarily the selective serotonin reuptake inhibitors (SSRIs) and of cognitive behavioral therapy (CBT). Medications and CBT rarely result in complete and lasting remission of symptoms, and residual symptoms are associated with a high rate of relapse. In most studies, a positive response is defined as a 30-50% improvement in symptoms and/or a global rating that the subject is much or very much improved. In adults, exercise has been used as a mono-therapy and as an augmentation therapy with antidepressant medication. Our recently completed randomized trial of exercise treatment in adults found response and remission rates of 46% and 42%, in those randomized to a public health dose of exercise. In adolescents, data on the use of exercise to treat MDD is relatively sparse. A 2006 Cochrane review of exercise to prevent and treat depression in adolescents found a small effect size in support of exercise, but the conclusion is based on evidence from a small number of randomized clinical trials of low methodological quality. In this exploratory R34, the specific aims of this application are to: 1) Develop a detailed Manual of Procedures (MOP) to conduct an acute-phase randomized trial of exercise to treat adolescent depression; 2) Develop estimates of recruitment yield from tests of various recruitment strategies; and, 3) Pilot test trial methodologies in (n=40) adolescents diagnosed with depression to ascertain estimates of treatment effect sizes, adherence and drop-out rates. To achieve these aims, the project is organized into 3 phases. Phase I will be the development of the first draft MOP that will adapt procedures developed from a previous trial examining two doses of exercise in treatment of adult MDD. Phase II will test specific recruitment methodologies to determine recruitment yields for each strategy and will pilot test screening procedures developed in Phase I. Phase III will be a pilot test of the intervention and will include development of baseline and outcome measures of exercise and depression; development and implementation of the experimental exercise treatment; and determination of the effects of exercise on depressive symptoms. Following the pilot study, we will finalize all procedures for the MOP and obtain estimates of effect sizes, adherence and drop out rates. These data will allow us to specify all study procedures necessary to meet standards of high methodological quality for a future, larger-scale, controlled study of exercise in depressed youth and will provide us with needed experience.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of DSM-IV Major Depression Disorder (MDD)
* Child Depression Rating Scale Revised > or = 40 at final screen
* 12 to 21 years of age
* On a stable dose of antidepressants or ADHD medication only
* Physically capable of exercise according to AHA and ACSM standards
* Able to pass illicit drug screen
* Perform < 20 minutes per day of moderate to vigorous physical activity
* Parental consent and participant assent
* Denver metropolitan area including Jefferson county

Exclusion Criteria:

* Chronic disease that would limit exercise
* Other psychiatric illness
* Suicidal or homicidal
* Concurrent psychotherapy
* Two previous failed SSRI trials or a failed trial of CBT
* Current pregnancy or breastfeeding

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Child Depression Rating Scale-Revised (CDRS-R) | repeated measures, 12-weeks

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | repeated measures, 12 weeks
The Multidimensional Anxiety Scale for Children (MASC) | baseline and 12 weeks
Adolescent Stress Questionnaire (ASQ) | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Dunn, PhD, Principal Investigator — Klein Buendel, Inc.